CLINICAL TRIAL: NCT05602935
Title: Efficacy and Safety of SOX Regimen Combined With Camrelizumab as Neoadjuvant Treatment in Locally Advanced Gastric Cancer: a Phase II, Single-arm Study
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Second Affiliated Hospital of Fujian Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEO-GASTRIC
Record Dates: First submitted 2022-10-24; First posted 2022-11-02 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2022-11

CONDITIONS: Stomach Neoplasms; Digestive System Neoplasms; Neoplasms; Digestive System Diseases; Stomach Diseases; Neoplasms by Site
Keywords: gastric cancer; neoadjuvant chemoimmunotherapy; neoadjuvant immunotherapy
MeSH Terms: conditions — Stomach Neoplasms; Digestive System Neoplasms; Neoplasms; Digestive System Diseases; Stomach Diseases; Neoplasms by Site | interventions — camrelizumab; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Camrelizumab+SOX (Experimental): The patients in the experimental arm will receive camrelizumab concurrently with SOX(S-1 and oxaliplatin).
  Interventions: Drug: Camrelizumab; Drug: SOX; Procedure: Surgery

INTERVENTIONS:
Drug: Camrelizumab — 200mg, intravenously, d1
Drug: SOX — SOX (S-1: 40~60mg, orally twice daily on days 1 to 14, oxaliplatin 130mg/m2 intravenously on day 1, 21 days per cycle)
Procedure: Surgery — Surgery

SUMMARY:
This is a single-arm, phase II study of camrelizumab combined with SOX regimen in subjects with resectable locally advanced gastric cancer. The patients will receive camrelizumab ,S-1 and oxaliplatin given every 3 weeks for 3 cycles as neoadjuvant therapy. After the surgery, adjuvant therapy which includes camrelizumab and SOX regimen will begin.

ELIGIBILITY:
Inclusion Criteria:

1. Age older than 18 years of age;
2. Histologically or cytological confirmed gastric or gastroesophageal junction adenocarcinoma;
3. Without prior systematic therapy;
4. The Eastern Cooperative Oncology Group Performance status (ECOG PS) 0-1;
5. With measurable lesions according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1;
6. Clinically diagnosed stage cT3-4bN1-3M0 evaluated by CT/MRI/EUS;
7. Life expectancy longer than 12 months;
8. Adequate function of blood, heart, liver, kidney and thyroid.

Exclusion Criteria:

1. History of immunodeficiency, including HIV positive, or other acquired or congenital immunodeficiency disease, or history of organ transplantation or allogeneic bone marrow transplantation;
2. Unresectable tumor evaluated by investigator;
3. Present of poorly controlled cardiac symptoms or disease, including but not limited to: (1) heart failure with NYHA class II or above (2) unstable angina, （3）myocardial infarction occurred within 1 year (4) clinical significance supraventricular or ventricular arrhythmias without clinical intervention or poorly controlled after clinical intervention;
4. With tumors in other sites;
5. History of any active autoimmune disease, including but not limited to: interstitial pneumonia, enteritis, hepatitis, hypohysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism (may be considered after hormone replacement therapy);Patients with psoriasis or childhood asthma/allergy who have been in complete remission and do not need any intervention as adults may be considered for inclusion, but patients requiring medical intervention with bronchodilators may not be included;
6. Has a history of allergy to monoclonal antibody, any component of PD-1 Inhibitor, S-1 and oxaliplatin;
7. With any mental illness;
8. Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2020-09-16 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete response (pCR) rate | 2-4 months
  The AJCC TRG system was used in this study to determine the effects of treatment. TRG 0 indicating athologic complete response (pCR)

SECONDARY OUTCOMES:
R0 resection rate | 2-4 months
Overall response rate(ORR) | 2-4 months
Disease control rate(DCR) | 2-4 months
Major pathological response (MPR) | 2-4 months
  The AJCC TRG system was used in this study to determine the effects of treatment.
Adverse events (AE) rate | 3 years
Event-free survival(EFS) | 3 years
Overall survival(OS) | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhong WJ, Lin JA, Wu CY, Wang J, Chen JX, Zheng H, Ye K. Efficacy and safety of camrelizumab combined with oxaliplatin and S-1 as neoadjuvant treatment in locally advanced gastric or gastroesophageal junction cancer: A phase II, single-arm study. Cancer Med. 2024 Feb;13(3):e7006. doi: 10.1002/cam4.7006. PMID 38400680